CLINICAL TRIAL: NCT05086640
Title: Evaluation of the Effectiveness of the Local Application of Lemon in the Prevention of Blisters in Ultra-trail Runners
Acronym: BS-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Formation et de Recherche en Médecine de Montagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Blisters-stop 2
Record Dates: First submitted 2021-09-03; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-05

CONDITIONS: Blister of Foot; Sport Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lemon foot (Experimental): Application of Lemon in the Prevention of Blisters on one feet
  Interventions: Other: Lemon foot to prevent blister
- Control foot without lemon (No Intervention): No application of Lemon or any other prevention cream in the Prevention of Blisters on one feet

INTERVENTIONS:
Other: Lemon foot to prevent blister — The investigators make the hypothesis that the local application of Lemon allows a reduction of the number of blisters on ultra-trail.
  Arms: Lemon foot

SUMMARY:
For more than a decade, worldwide participation in ultra-marathons and ultra-trails (running races longer than the 42.195 km marathon) has been increasing. Although considered benign, blisters are a common problem, with serious consequences and limiting performance.

Although blisters are a major factor limiting endurance performance, they are a reason for only 5.8% of ultra-trail runners to quit.

While equipment is improving and participants are increasing and intensifying their training, there is no consensus on the prevention of blisters in ultra-trail running, even though it is the number one factor limiting sports performance. There are few prospective interventional studies on the prevention of blisters during outdoor activities.

On many running forums, there is the hypothesis that lemon applied to the feet prevents the appearance of blisters. This hypothesis has never been scientifically studied.

The investigators hypothesize that the local application of Lemon allows a reduction in the number of blisters on ultra-trail.

The objective of this Blisters-stop 2 study is to evaluate the efficacy of local application of Lemon in preventing the appearance of blisters.

DETAILED DESCRIPTION:
The patients included will be runners registered in a trail of a distance greater than 40km for whom Lemon will be applied on the friction zones of one foot as a preventive measure (28 days).

The study is coordinated by IFREMMONT and the Pays du Mont Blanc Hospitals and 82 patients must be included in order to obtain statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Ultra-trail participants with validated registration
* Major (≥ 18 years old)

Exclusion Criteria:

* Presence of blisters or other skin lesions on the feet 28 days before the race
* Amputation of one or two feet
* Allergy to lemon
* Psychiatric disorders making comprehension impossible
* Lack of social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence or not of blisters at the end of the ultra-trail or at the time of abandonment. | up to 1 week
  Blisters on each feet or non

SECONDARY OUTCOMES:
Feasibility of the protocole | up to 1 week
  Easy to follow for runners, lemon used every day, how mutch misses
Compliance | up to 1 week
  Compliance to the protocole
Tolerance | up to 1 week
  Tolerance to the protocole
Main locations of residual blisters | up to 1 week
  Where on each feet
Severity of residual blisters | up to 1 week
  Severity

CONTACTS AND LOCATIONS:
Overall Officials: Corentin Tanné, Principal Investigator — Institut de Formation et de Recherche en Médecine de Montagne
Locations (1):
- Ifremmont, Chamonix, France

IPD SHARING:
Plan to Share IPD: No